CLINICAL TRIAL: NCT01997138
Title: Effects of Intraarticular IL1-Ra on Pain and Inflammatory Mediators After Knee Arhroscopy -a Double Blind, Placebo Controlled Study Using Microdialysis Technique
Brief Title: Effects of Intraarticular IL1-Ra on Pain and Inflammatory Mediators After Knee Arhroscopy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Too few recruitable patients
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other); Lovisenberg Diakonale Hospital (Other)
Responsible Party: Principal Investigator, Leiv Arne Rosseland, Professor MD, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: anakinrapain1
Record Dates: First submitted 2013-11-22; First posted 2013-11-27 (Estimated); Last update posted 2021-06-11 (Actual); Status verified 2021-06

CONDITIONS: Knee Injuries
Keywords: pain, inflammation, surgery
MeSH Terms: conditions — Knee Injuries; Pain; Inflammation | interventions — Interleukin 1 Receptor Antagonist Protein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anakinra (Experimental): Anakinra 100 mg in 2 ml saline IA
  Interventions: Drug: Anakinra 100 mg in 2 ml saline IA
- Placebo (Placebo Comparator): Saline 2 ml IA
  Interventions: Drug: Anakinra 100 mg in 2 ml saline IA

INTERVENTIONS:
Drug: Anakinra 100 mg in 2 ml saline IA
  Other Names: Kineret

SUMMARY:
This project investigates the relation between acute pain and local inflammation. Pain reported by the patients for knee arthroscopy are compared with local changes in inflammatory mediators by using microdialysis technique. Patients with moderate-to-severe pain are included in a randomized placebo-controlled trial of anakinra given intra-articularly.

DETAILED DESCRIPTION:
The effects of the recombinant IL-1 receptor antagonist anakinra both on acute pain and post operative inflammation will be evaluated. On inclusion, pain intensity will be measured on a five-point verbal rating scale (0= no pain, 1=mild pain, 2=moderate pain, 3=severe pain, and 4=intolerable pain), and on a visual analogue scale (0-100mm). VAS scale will be repeated at 20, 40, 60, 80, 100, 120, 140, 160, 180 and 200 minutes after inclusion / intervention. The patients will also rate pain intensity during a 5 meters walk at 200 minutes (evoked pain). The patient will rate pain at rest and evoked pain 24, 48 and 72 h after intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Otherwise healthy patients (ASA 1 and 2) undergoing knee arthroscopy in general anaesthesia.
2. Being informed about and willing to participate in the study -

Exclusion Criteria:

1. Pregnancy or lactation. Fertile women will be asked if they may be pregnant, and offered a pregnancy test if there is doubt.
2. Established osteoarthritis or synovitis
3. Known intolerance to anakinra
4. Kidney failure (Creatinine clearance <30ml/min)
5. History of frequent infectious diseases or immunodeficiency
6. Heart failure
7. History of drug -or alcohol abuse
8. Participation in other synchronous clinical trials
9. Perioperative steroid treatment, perioperative paracetamol (12 hrs), NSAIDs (24 hrs) or COX2-inhibitors (48 hrs).
10. Use of tourniquet for bloodless field
11. Strong preoperative pain (VRS ≥3)
12. Intolerable postoperative pain (VRS=4)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03; Primary Completion 2018-01 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Pain relief | 72h
  Selv reported pain

SECONDARY OUTCOMES:
Resuce analgesic drug consumption | 72h
  Need for and consumption of resuce analgesic drug

OTHER OUTCOMES:
Side effects | 72h
  Selv reported side effect according to CRF

CONTACTS AND LOCATIONS:
Locations (1):
- Lovisenberg Diakonal Hospital, Oslo, Norway